CLINICAL TRIAL: NCT07376356
Title: A Randomized Controlled Trial of Executive Function Intervention for Children With Autism Spectrum Disorder(ASD) Combining Digital Application and Parent Coaching
Brief Title: Executive Function Intervention for Children With ASD Combining a Digital App and Parent Coaching
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, So Hyun Kim, Associate Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2025-0286; 00209635 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Waitlist Control Group Design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChuckChuck Step Intervention (Experimental): Children will participate in an executive function training intervention delivered via a digital application provided by Neudive. The intervention consists of daily(Mon-Fri) child-friendly and school-context games that lasts approximately 15 minutes for six weeks. Meanwhile, parents will participate in a parent mediated executive function intervention delivered via telehealth over six weekly 60 minute group sessions. Sessions will include psychoeducation, delivering of executive function related strategies, and interactive activities to promote engagement and skill practice. This program is designed to train children with Autism Spectrum Disorder in executive function and support parents of those children through parent mediated intervention.
  Interventions: Behavioral: ChuckChuck Step
- Waitlist Control (Active Comparator): After collecting data for all timepoints, children in the waitlist control group will participate in the same EF(Executive Function) training intervention delivered via a digital application provided by Neudive. Meanwhile, parents will participate in an abbreviated parent mediated EF intervention delivered via telehealth over three weekly 60 minute group sessions. Sessions will consist of the same contents as the intervention group, including psychoeducation, delivering of EF related strategies, and interactive activities to promote engagement and skill practice.
  Interventions: Behavioral: ChuckChuck Step (Shortened Parent Coaching)

INTERVENTIONS:
Behavioral: ChuckChuck Step — Our intervention will consist of a daily(Mon-Fri), six-week, digital application based intervention (15 minutes per day) for children and six-week telehealth based group intervention (60 minutes per week) to support both children with ASD (5- to 8-year-olds) and their parents regarding executive function hardships. This program provides training for inhibition, working memory, planning and organizing, cognitive flexibility, and emotion regulation. Children will practice these aspects of executive function while playing child-friendly games with the storyline being based on everyday school related themes. Games will consist of go-nogo tasks, following arrows, memory games etc. Parents will learn about these aspects of executive function through real-time telehealth and will be provided with strategies to further promote growth of executive function abilities in their children. The parent mediated intervention curriculum moves beyond didactic instruction by combining psychoeducation with
  Arms: ChuckChuck Step Intervention
Behavioral: ChuckChuck Step (Shortened Parent Coaching) — Children in the waitlist control group will receive the same intervention as the intervention group after the waitlist period.
  Parents in the waitlist control group will receive an abbreviated version(three-week) of the parent mediated intervention with the same contents as the intervention group.
  Arms: Waitlist Control

SUMMARY:
The purpose of this randomized controlled study is to develop and evaluate a digital cognitive control intervention that integrates a digital application-based child training program with an online parent coaching program for early school-aged children aged 5-8 with autism spectrum disorder (ASD) and their caregivers in South Korea. This intervention is designed to enhance clinical applicability, sustainability, and generalization to daily life of executive skills through active parental involvement. This study has three primary aims: (1) to examine the feasibility, acceptability, and implementation fidelity of the integrated child-parent digital intervention, (2) to investigate the effects of the intervention on children's cognitive control and executive function using behavioral assessments and neurophysiological measures (e.g., EEG), as well as on parents' use of cognitive control-supportive strategies in daily contexts, and (3) to assess whether intervention related changes generalize to real-world functioning, including children's adaptive behavior, academic readiness, and social functioning, as reported by parents, and whether these effects are maintained over time.

DETAILED DESCRIPTION:
Early school-aged children with autism spectrum disorder (ASD) frequently experience difficulties in executive functioning, including challenges in inhibitory control, working memory, cognitive flexibility, planning, and emotion regulation. These skills are essential for successful adaptation to school environments, peer relationships, and daily routines, and early deficits have been shown to predict long-term outcomes related to academic achievement, social participation, independent living, and mental health. Despite their clinical importance, there remains a lack of developmentally appropriate, evidence-based executive functioning interventions tailored for early school-aged children with ASD.

Parent-mediated interventions have demonstrated effectiveness in improving children's cognitive control and reducing problem behaviors, particularly due to their strength in promoting generalization of skills to everyday contexts such as home and school. However, these interventions are often limited by caregiver burden, parenting stress, and difficulties maintaining consistency and long-term adherence. In contrast, child-focused digital interventions provide structured, engaging, and algorithm-based training but frequently show limited generalization beyond the intervention setting. Integrating child-centered digital cognitive control training with structured parent coaching may therefore address the limitations of each approach and yield a more effective and sustainable intervention model.

The purpose of this randomized controlled study is to develop and evaluate a digital cognitive control intervention that integrates a digital application-based, game-oriented child training program with an online parent group coaching program for children aged 5 to 8 years with ASD and their caregivers in South Korea. The intervention targets core components of executive functioning within everyday school-related contexts and aims to enhance caregivers' understanding of executive functioning, their capacity to scaffold and reinforce skills in daily life, and the generalization of intervention gains beyond the digital environment, particularly for high-functioning children with ASD who have limited access to specialized services.

A total of 40 children with ASD (aged 5 years 0 months to 8 years 11 months) and their primary caregivers will be recruited in South Korea. Eligible children must meet DSM-5 or Autism Diagnostic Observation Schedule criteria, demonstrate phrase-level expressive language (ADOS modules 2 or 3), and have a nonverbal IQ of 70 or above. Participants will be randomly assigned to either an intervention group (n=20) or an active control group (n=20) using stratified block randomization based on age, sex, and nonverbal IQ. Children in both groups will complete a six-week home-based digital application cognitive control training program conducted five days per week for approximately 15 minutes per session. In addition, caregivers in the intervention group will participate in a six-week online parent group coaching program with weekly 60-minute sessions, while caregivers in the active control group will receive a shortened parent coaching program after their assessment period. Outcomes will be assessed at three time points using behavioral tasks, parent-report measures, and electroencephalography (EEG) to provide a comprehensive evaluation of intervention efficacy and underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Children in South Korea aged 5-8
* Children with previous medical diagnosis of ASD or children categorized as "Autism" or "Autism Spectrum" after administering ADOS-2
* Children with language abilities that meet the eligibility for ADOS-2 Module 2 or 3
* Children with cognitive functioning assessed using the Wechsler Preschool and Primary Scale of Intelligence and a nonverbal IQ of 70 or above

Exclusion Criteria:

* Children with significant intellectual disability
* Children with significant language delay

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
EF Touch | baseline, immediately after the intervention, 6-weeks follow-up
  EF Touch is a child-friendly computerized EF task, administered on a touch-screen tablet. The use of EF Touch will allow us to target fine-grained, multiple EF domains, including inhibitory control ("Spatial Conflict Arrows"), working memory ("Pick the Picture"), and attention shifting ("Something's the Same). The proportion of correct trials for each domain will be used as an outcome.
HTKS | baseline, immediately after the intervention, 6-weeks follow-up
  HTKS is a tool that measures behavioral self-regulation in children and consists of short tasks suitable for children 4-8 years of age. The game consists of up to four behavioral rules, and the examiner elicits a natural response from the child, such as "touch your head" or "touch your knee," and then switches the rules in a "reverse" fashion (e.g., "Now touch your toes when I tell you to touch your head"). This should take about 5 minutes.
Stroop | baseline, immediately after the intervention, 6-weeks follow-up
  The Stroop Color and Word Test Children's Version is a tool for measuring the efficiency of inhibitory control, and the Korean version of the test was standardized for reliability and validity in 2006. During the test, words that do not match in color and letter are presented, and the subject must respond to the color instead of the letter, which is an automatic response. It is a neuropsychological test suitable for ages 5-14 and takes about 5-10 minutes.
ACE | baseline, immediately after the intervention, 6-weeks follow-up
  The ADHD Comprehensive Evaluation (ACE) is a standardized, multi-component assessment tool designed to provide a comprehensive evaluation of ADHD-related functional impairments as well as core components of cognitive control. The ACE includes the Korean Attention Test (KAT), the Korean ADHD Rating Scale-5 (K-ARS-5), a Working Memory Test (WMT), and an Executive Function Test (Computerized Trail Making Test; C-TMT). It is a neuropsychological assessment battery suitable for children aged 5 to 15 years and assesses key domains of attention, working memory, and executive functioning relevant to cognitive control. WMT and C-TMT will be utilized in this study and each component requires approximately 5 to 15 minutes to administer.
BRIEF | baseline, immediately after the intervention, 6-weeks follow-up
  The Korean Behavior Rating Inventory of Executive Function is a standardized parent report to observe children's cognitive control. It assesses behavior in executive functioning and is used to assess children with learning disabilities and attention disorders, as well as neurological, psychiatric, and medical conditions. It includes 86 items measuring various aspects of each executive function, which are categorized into eight clinical scales and two validity scales to provide a balanced view of the child's behavior. The test is intended for children ages 5-18 and takes approximately 15 minutes to complete.
EDI | baseline, immediately after the intervention, 6-weeks follow-up
  The Emotion Dysregulation Inventory is an informant questionnaire that assesses emotion regulation difficulties. It consists of 30 items, and informants (parents/caregivers) rate each item (e.g., "has sudden outbursts of emotion," "doesn't seem to enjoy anything") on a 5-point Likert scale ranging from "not at all" to "very severe" based on their observations of the child's functioning over the past 7 days.
Intervention feasibility and acceptability survey | immediately after the intervention
  Intervention feasibility and acceptability survey will be systematically evaluated using multiple indicators relevant to clinical trial implementation. Intervention feasibility will be assessed by tracking enrollment and retention rates across key demographic characteristics, the proportion of participants deemed ineligible based on screening procedures and clinical assessments, and data acquisition rates for cognitive control-related tasks administered before and after the intervention. Intervention acceptability will be evaluated using Likert-scale ratings and open-ended questions to capture participants' experiences and perceptions of the program (e.g., "Please describe the strengths of the intervention program," "Please describe any difficulties you experienced while participating in the intervention").

SECONDARY OUTCOMES:
Vineland | baseline, immediately after the intervention, 6-weeks follow-up
  The Vineland Adaptive Behavior Scale is a standardized parent report to measure children's social skills, communication, and adaptive behavior. It can be administered on children 0 to 90 years of age and consists of 433 items, each scored on a 0, 1, or 2-point scale. It provides measures of overall adaptive behavioral functioning and subdomains of adaptive behavior (communication, life skills, social, and motor skills).
K-WFA | baseline, immediately after the intervention, 6-weeks follow-up
  The Korean Wechsler Fundamentals: Academic Skills is a brief, standardized achievement assessment adapted and normed from the original Wechsler Fundamentals: Academic Skills (WFA) to evaluate core academic skills essential for learning in educational settings. In the present study, the K-WFA will be used to assess children's academic skill levels and changes associated with intervention effects. The measure evaluates fundamental domains including word reading, reading comprehension, writing, and numerical calculation. The K-WFA consists of parallel forms (Form A and Form B), allowing for pre- and post-intervention assessment, and enables rapid evaluation of functional academic skills as well as monitoring of learning-related changes over time.
PIPPS | baseline, immediately after the intervention, 6-weeks follow-up
  The Penn Interactive Peer Play Scale is a play behavior assessment developed to understand children's interactions with peers and to be consistently rated by parents or teachers across settings during early childhood. Our study will utilize the parent report to assess children's play in home and neighborhood environments. The parent report records the level of frequency at which each behavior was observed during the child's free play over a 2-month period. It consists of 32 4-point Likert scales and results include the following domains: play disruption, play interaction, and play disengagement.
CBCL | baseline, immediately after the intervention, 6-weeks follow-up
  The Child Behavior Checklist is a standardized parent-report measure used to assess children's emotional and behavioral problems, with age-specific versions to ensure developmental appropriateness. In this study, it will be administered based on the child's age: the CBCL 1.5-5 will be used for children aged 18 months to 5 years, and the Korean Child Behavior Checklist for Ages 6-18 (K-CBCL 6-18) will be used for children aged 6 to 18 years. The Korean CBCL 1.5-5, published in 2008, includes a Problem Behavior Scale and a Language Development Scale, with the problem behavior items assessing internalizing and externalizing difficulties as well as DSM-oriented symptom domains using a 3-point Likert scale. The K-CBCL 6-18, released in 2010 following nationwide standardization, consists of a 113-item, 3-point Likert-scale Problem Behavior Scale that captures a broad range of emotional and behavioral functioning based on parent report.
BOSCC | baseline, immediately after the intervention, 6-weeks follow-up
  The Brief Observation of Social Communication Change is a behavioral observation tool originally developed to measure pre- and post-intervention treatment effects in children with autism. The first 5-6 minutes (Segment A) and the second 5-6 minutes (Segment B) of free play between an interventionist or caregiver and a child with autism are filmed. The number and quality of the child's social communication and interactions (e.g., eye contact, facial expressions, gestures, social cues and responses) and limited and repetitive interests or behaviors (e.g., sensory-seeking behaviors) are observed between 10 and 15 minutes.
EEG | baseline, immediately after the intervention, 6-weeks follow-up
  We found that EEG central prefrontal theta oscillations, measured using time frequency analysis, provide a new window into understanding the neural basis of cognitive control in children with autism. Children with ASD between ages of 5-6 years showed higher theta power while producing incorrect responses, which require more brain resources than correct responses during go/no-go cognitive tasks. This was correlated with better performance on behavioral cognitive control tasks. In this study, we plan to measure error-related theta oscillations and error-related negativity (ERN) using EEG tasks. We will use the Zoo Game, a validated EEG task that is developmentally appropriate for children. It is a go/no-go task designed to optimize child engagement and motivation by combining animal pictures and an engaging story to make the go and no-go clear and easy for children to understand, and has been shown in previous research to be suitable for children with autism.
K-PSI | baseline, immediately after the intervention, 6-weeks follow-up
  The Korean Parenting Stress Index-Fourth Edition Short Form (K-PSI-4-SF) is a parent self-report measure with items extracted from the K-PSI-4 that are most sensitive for measuring parenting stressors. It consists of three subscales (Parental Distress, Parent-Child Dysfunctional Interaction, and Demanding Child) that assess parent characteristics, parent-child interactions, and parent-perceived child characteristics that influence parenting stress, with 12 items per scale. Items are rated on a 5-point Likert scale with varying anchor statements (e.g., from "strongly disagree" (1) to "strongly agree" (5); from "definitely not adequate as a parent" (1) to "a very good parent" (5); and from "much easier than expected" (1) to "much more difficult than expected" (5)). Total scores range from 36 to 180, with higher total scores indicating greater levels of stress experienced in parenting.
BDEFS | baseline, immediately after the intervention, 6-weeks follow-up
  The Barkley Deficits in Executive Functioning Scale, which was developed to assess executive function deficits in adult ADHD patients, consists of 89 items with five subdomains: 'Self-management of time', 'Self-organization/problem solving', 'Self-control', 'Self-motivation', and 'Self-regulation of emotions', measured with a 4-point Likert scale. In this study, we will use the Korean version of Short Form (K-BDEFS-SF) to assess the presence of executive function and ADHD symptoms in daily lives of caregivers of children with autism.
ERQ | baseline, immediately after the intervention, 6-weeks follow-up
  This study will use the 10-item Emotion Regulation Questionnaire to measure how parents experience and express their emotions, i.e., how they cognitively interpret and regulate emotion in their daily lives as caregivers. Each item is rated on a 7-point Likert scale from "not at all" to "very much so" (e.g., "When I want to feel more positive, I change the way I think about the situation," "I suppress my emotions.").
Loneliness and Social Isolation Scale | baseline, immediately after the intervention, 6-weeks follow-up
  The Loneliness and Social Isolation Scale is an instrument that encompasses both objectively measurable "social network" and an individual's subjective perceptions of "social support" and "loneliness" to estimate the complex concept of "social isolation". It consists of 6 questions and is self-reported. Each item is scored on a 0-3 scale.
UCLA Loneliness Scale | baseline, immediately after the intervention, 6-weeks follow-up
  The UCLA Loneliness Scale was developed by Russell et al. in 1978 and has been the most widely used instrument in loneliness research both domestically and internationally. Based on the definition of Weiss (1973), it defines loneliness as 'a state of extreme distress due to relational deficiency'. The revised version consists of 20 items, such as "I have no one to turn to", and each item is rated on a 4-point Likert scale ranging from "Not at all (1)" to "Often (4)." Higher scores indicate higher levels or frequency of loneliness. This study will use the Korean version of the UCLA Loneliness Scale, which is shortened to 8 items instead of the full 20-item scale.
Parenting Sense of Competence (PSOC) | baseline, immediately after the intervention, 6-weeks follow-up
  The Parenting Sense of Competence (PSOC) scale is a parent self-report measure used to assess parenting satisfaction and efficacy. Items are rated on a 6-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (6), with reverse-scored items included. Higher total scores indicate greater parental efficacy. Scores of 58 or below are interpreted as low, scores between 58 and 74 as average, and scores of 75 or above as high.
Parent Satisfaction Scale (PSS) | baseline, immediately after the intervention, 6-weeks follow-up
  The Parent Satisfaction Scale (PSS) is an instrument that assesses caregivers' subjective evaluation of their performance in the parenting role, as well as the positive and negative emotions arising from their parenting experiences. Items are rated on a 4-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (4), with reverse-scored items included. Higher total scores indicate greater satisfaction with the parenting role.
Autism Stigma and Knowledge Questionnaire (ASK-Q-2) | baseline, immediately after the intervention, 6-weeks follow-up
  The Autism Stigma and Knowledge Questionnaire (ASK-Q-2) will be used to assess caregivers' knowledge of and stigma toward autism. Items are scored dichotomously (agree = 1, disagree = 0).
National Institute for Special Education-Basic Academic Competence Tests | baseline, immediately after the intervention, 6-weeks follow-up
  The NISE tests will assess basic learning skills, such as reading and math, for students (ages 5 to 14).